CLINICAL TRIAL: NCT00239993
Title: An Open-Label, Randomized, Single Cross-over Study of Warm Compress Versus Usual Injection Site Preparation on Local Injection Site Reactions Among Persons With MS Who Perform Daily Injections of Copaxone®.
Brief Title: A Study to Evaluate the Impact of Using Warm Compress Prior to Daily Injections of Copaxone®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Neuroscience, Inc. (Industry)
Responsible Party: Thomas Smith, M.D., Vice President, Medical Affairs, Teva Neuroscience
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PM016
Record Dates: First submitted 2005-09-22; First posted 2005-10-17 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): skin reactions with the use of warm compress prior to performing a Copaxone® injection
  Interventions: Drug: glatiramer acetate
- 2 (Experimental): skin reactions without the use of warm compress prior to performing a Copaxone® injection
  Interventions: Procedure: Warm compress prior to injection of glatiramer acetate

INTERVENTIONS:
Drug: glatiramer acetate
  Other Names: Copaxone
  Arms: 1
Procedure: Warm compress prior to injection of glatiramer acetate
  Other Names: Copaxone
  Arms: 2

SUMMARY:
This study is designed to compare skin reactions with or without the use of warm compress prior to performing a Copaxone® injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years or older, with a diagnosis of RRMS
2. Willing and able to complete all procedures and evaluations related to the study.
3. Willing to provide Informed Consent

Exclusion Criteria:

1. Taking any other immunomodulatory therapy in conjunction with Copaxone®.
2. Has a significant medical illness other than MS which may interfere with the assessment of endpoints or the subject's participation in the trial for the full duration of the study.
3. Any situation which the investigator or nurse feels may interfere with participation in the study.
4. Pregnant, or trying to become pregnant, or breast feeding during the study.
5. Previously participated in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-08; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The number of local injection site reactions (LISRs) noted at 5-minutes post-injection | 2-week diaries kept by the patients for Period 1 and for Period 2

SECONDARY OUTCOMES:
The total and partial number of LISRs noted at 2-minutes post-injection The total and partial number of LISRs noted immediately after injection | 2-week diaries kept by the patients for Period 1 and for Period 2

CONTACTS AND LOCATIONS:
Overall Officials: MerriKay Oleen-Burkey, Ph.D, Study Director — Teva Neuroscience, Inc.
Locations (6):
- United States (6):
  - Fullerton Neurology & Headache Center, Fullerton, California
  - Neurological Center of South Florida, Miami, Florida
  - Springfield Neurology Associates, Springfield, Massachusetts
  - Multiple Sclerosis Care Center, Brooklyn, New York
  - Advanced Neurosciences Institute, Nashville, Tennessee
  - Virginia Beach Neurology, Virginia Beach, Virginia